CLINICAL TRIAL: NCT03831919
Title: Randomised Controlled Trial of Hoya SYNC III Design Lenses
Brief Title: Trial of Hoya SYNC III Design Lenses
Acronym: SYNCIII
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Institute of Optometry, London (Other)
Collaborators: University of Alicante (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SYNCIII
Record Dates: First submitted 2019-01-23; First posted 2019-02-06 (Actual); Last update posted 2020-07-30 (Actual); Status verified 2020-07

CONDITIONS: Computer Vision Syndrome
Keywords: ocular accommodation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- SYNC III accommodative support lenses (Experimental): Wear spectacles with SYNC III accommodative support lenses (add +0.75)
  Interventions: Device: SYNC III
- control (Placebo Comparator): Wear single vision spectacles (no add)
  Interventions: Device: single vision lenses

INTERVENTIONS:
Device: SYNC III — Hoya SYNC III design spectacle lenses
  Arms: SYNC III accommodative support lenses
Device: single vision lenses — single vision spectacle lenses with no addition
  Arms: control

SUMMARY:
Many people using computers or digital devices (e.g., smartphones or tablets) experience eyestrain and this has been called Computer Vision Syndrome (CVS) or Digital Eye Strain. Spectacle lens manufacturers have designed products to alleviate the symptoms of CVS. One such product, designed by Hoya (SYNC III), aims to do this by providing accommodative support. The present study is a parallel group double-masked RCT of people with CVS. One group will receive Hoya SYNC III lenses and the other (control) group single vision (SV) lenses. The main aims are to evaluate whether:

1. binocular vision and accommodative functions at baseline can predict participants who benefit from SYNC III design lenses;
2. the wearing of SYNC III design lenses is associated with any changes in binocular and accommodative functions at 6 months of follow-up;
3. the wearing of lenses with accommodative support reduce the symptoms of computer vision syndrome at 3 and 6 months of follow-up.

Participants will be examined three times: at baseline and three and six months after receiving their lenses. The group who receive control lenses will be provided with SYNC III lenses at the end of the six month trial for a brief one week follow-up evaluation.

DETAILED DESCRIPTION:
Background Aims

The aims of the research are to use a parallel group randomised controlled trial to:

1. Evaluate whether binocular vision and accommodative functions at baseline can predict any participants who benefit from SYNC III design lenses;
2. Evaluate whether the wearing of SYNC III design lenses is associated with any changes in binocular and accommodative functions at 6 months of follow-up;
3. Evaluate whether the wearing of lenses with accommodative support may reduce the symptoms of computer vision syndrome at 3 and 6 months of follow-up.

Methods Design The research is a double-masked randomised controlled trial. Participants will be randomly allocated to two groups, one of whom wears SYNC III design lenses and the other who will wear SV control lenses.

The research involves thirty participants (15 wearing SYNC III design and 15 with SV) who will be seen at the Institute of Optometry, London; and 60 participants (30 wearing SYNC III design and 30 with SV) seen at the University of Alicante.

Procedure The research has received approval from the REC of the Institute of Optometry.

Potential participants will be sought from workplaces and free advertisements in London. Potential participants will initially be contacted by telephone or email to see if they meet the entry criteria. Those who do will be invited to complete the CVS-Q and return this to the researcher to determine if they meet selection criterion described later. Those that do will be invited to participate in the research and will be sent full information and a consent form and given the opportunity to have any questions answered. For those that wish to proceed, an appointment will be arranged for the baseline assessment and they will be asked to bring their consent form to that appointment, as well as any optical spectacles that they usually wear.

The baseline assessment will start with the consent process and attendees will be given the opportunity of having any further questions answered before they sign the consent form. The baseline assessment will only proceed if participants sign the consent form.

Prior to the baseline assessment, participants will have already completed and returned the CVS-Q. The researcher will check the response with the participant and record the results.

During the baseline assessment in the unlikely event that any pathology is detected that requires medical attention then the participant will be referred according to local protocols and excluded from the research study (a note of the number of participants, if any, excluded in this way will be kept). All participants who are not excluded because of pathology will be allocated a research ID number.

Hoya will supply the research centres with sample spectacle frames. At the end of the baseline assessment, participants will choose a frame that they are happy to wear and which the researcher considers fits properly. The fitting parameters will be measured with the Hoya VisuReal instrument, which will be provided by Hoya.

The participant ID number, new spectacle prescription, frame choice, and fitting parameters will be sent to BE. BE will keep a confidential table of pre-determined (using a random number generator) random allocation codes which will determine whether, for example, participant 01 will receive the SYNC III design lenses or SV control lenses (there is a random 50:50 chance of each intervention for each participant). BE will add this information to the other information he receives from the research centre and will send this to Hoya Lens Iberia in Madrid who will manufacture the spectacles for each participant and return these to the research teams. There will be no markings on the lenses and the research centres will not investigate the lenses to see if they are SYNC III design or SV. The research centres will arrange an appointment for the participant to collect the spectacles and will arrange follow-up appointments after approximately three and six months.

At the collection appointment the fit of the spectacles will be checked and adjusted if required. The distance and near visual acuities will be checked to ensure they are as expected. The participant will be instructed to wear the spectacles for all work with digital devices and to contact the local research team if there is any difficulty complying with this instruction.

Approximately once a month a member of the local research team will telephone or email each participant to remind them to wear their spectacles, and to remind them of the date of their next appointment.

At the three months and six months follow up appointments the tests in Table 2 will be repeated (except for ophthalmoscopy and biomicroscopy). For all these tests (except ocular motility), the participant will wear the same refractive correction as worn at the baseline assessment. This is to facilitate the detection of any changes from the baseline accommodative and binocular function that may be attributable to wearing SYNC III design lenses. When the participant completes the CVS-Q, they will be asked to do so considering the symptoms they have experienced (if any) with the research spectacles they have been wearing.

At the end of the final appointment (after six months of wear), after all the tests have been completed, the researcher will inspect the lenses in the research spectacles to see if they are SYNC III design or SV. They will inform the participant and, if they have been wearing SYNC III design, the participant will be allowed to keep the spectacles.

Participants who have been wearing control SV lenses will be offered SYNC III design lenses (this will be made clear in the study information that is given to potential participants before recruitment, to encourage participation). These SYNC III design lenses will be sent to participants (in identical frames but with a white mark on the inside of the right side) after the six months appointment, via the research team. Once these have been worn for one week, the researcher will telephone the participant to explore their experience with these lenses compared with the SV control lenses. Participants will be asked, if they could keep only one pair, whether they would prefer the SYNC III design or the SV controls. They will, however, be permitted to keep both pairs. It is considered that allowing these participants to keep two pairs of frames will be a worthwhile gesture to thank participants who have worn SV lenses for six months.

It should be noted that this is not a formal cross-over trial, but rather the participants who received SV lenses throughout the main trial will receive SYNC III spectacles for just one week. A full cross-over trial is considered to be impractical because the six months period with each intervention (which is necessary to determine any effect of SYNC III design on accommodation) would make a full cross-over trial prohibitively lengthy.

Details Interventions SYNC III accommodative support lenses are manufactured by Hoya with three accommodative support "boost" powers, +0.57, +0.95, +1.32. A sister company, Seiko, also use the SYNC III design but with different accommodative support powers, including +0.75. A recent research study compared accommodative support from +0.50, +0.75, and +1.25 and found +0.75 to be the preferred option for most participants. Therefore, a SYNC III design with +0.75 accommodative support will be used in the present research.

The control lenses will be standard Hoya single vision aspheric lenses. Both the experimental and control lenses will be made from 1.6 refractive index plastic lenses with a standard anti-reflection coating, and neither will have blue-blocking coatings.

Attrition The study will follow an "intention to treat" principle. It is considered inevitable that some participants will drop out during the trial, and no new participants will be started in their place.

Analyses

1. An Excel spreadsheet will be developed for recording results.
2. Data will be entered in the Excel spreadsheet and analysed using Excel and SPSS.
3. Each variable (see Table 2) will be tested using the Shapiro-Wilk test for normality and parametric and non-parametric statistics will be used as appropriate.
4. ANOVA will be used to determine whether the CVS-Q scores at three and six months differ from those at baseline and to test the effect of the intervention worn.
5. Similarly, ANOVA will be used to determine whether there is any change on the accommodative or binocular vision variables with each intervention after three and six months.
6. Multivariate analysis will be carried out to evaluate the association between variables and control the confounding factors

Dissemination Regardless of the outcome, the results of the study will be submitted for publication in a peer-reviewed journal. The work will also be available for presentation at the Hoya International/KOL meeting and may also be submitted for presentation at scientific and clinical conferences, with the agreement of all the researchers.

Ethical considerations The research will conform to the tenets of the Declaration of Helsinki. Personal data will only be used to contact participants and will be stored on a separate password protected spreadsheet to the research data. This will be stored securely at the IoO and at the University of Alicante.

Participants will only start the trial once they have signed a consent form. Participants will be free to withdraw at any time. If they do withdraw then they will be invited to give a reason, but it will be made clear that they do not have to give a reason. If they withdraw they will be entitled to keep any spectacles that have been supplied.

The participant information sheet will make clear to participants that they will not be receiving an NHS sight test or optical prescription. At the end of the research, upon request the participant will be given a written copy of the specification of the spectacles they have worn in the research to show to their optometrist. Participants will be told that the research does not replace the need for regular eyecare with a community optometrist.

The research, data entry, analyses, and writing-up will be carried out independently of Hoya. The work will be disseminated, as outlined above, regardless of the outcome. Publications and presentations will acknowledge the funding support but will make it clear that the research and dissemination was carried out independently of Hoya who will have no say in the content of publications.

ELIGIBILITY:
Inclusion Criteria:

1. Aged between 18 and 40 years;
2. In a typical working day, spends at least 2 hours viewing digital devices (e.g., desktop, laptop, tablet, smart phone);
3. Symptoms associated with the use of digital devices, quantified as a score of six points or more on the CVS-Q questionnaire instrument;1
4. Use of spectacles, at least 6, months previous to the beginning of the study;
5. Refractive error between +6.00 to -8.00 with cyl up to 4.00DC.

Exclusion Criteria:

1. Previous use of accommodative support lenses
2. Ocular pathology requiring referral to an ophthalmologist
3. Wears contact lenses when using computers
4. Strabismus

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2019-01-07 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Change in CVS-Q | Baseline, three-month follow-up, six-month follow-up
  Computer vision syndrome quality of life instrument
Change in heterophoria | Baseline, three-month follow-up, six-month follow-up
  Dissociated heterophoria using Prentice test.
Change in aligning prism | Baseline, three-month follow-up, six-month follow-up
  Associated heterophoria using Mallett unit
Change in near point of convergence | Baseline, three-month follow-up, six-month follow-up
  NPC, push-up
Change in amplitude of accommodation | Baseline, three-month follow-up, six-month follow-up
  push-up
Change in accommodative lag | Baseline, three-month follow-up, six-month follow-up
  MEM retinoscopy
Change in accommodative facility | Baseline, three-month follow-up, six-month follow-up
  +-1.50 flippers

SECONDARY OUTCOMES:
Fusional reserves | Baseline, three-month follow-up, six-month follow-up
  near
Stereopsis | Baseline, three-month follow-up, six-month follow-up
  EyeGenius

CONTACTS AND LOCATIONS:
Overall Officials: Bruce Evans, PhD, Study Director — Institute of Optometry
Locations (2):
- University of Alicante, Alicante, Spain
- Institute of Optometry, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
the plan is to share anonymised data
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: within 1 year of end of study for unspecified period
Access Criteria: Genuine requests from researchers Only anonymised data will be provided

REFERENCES:
- [Background] Segui Mdel M, Cabrero-Garcia J, Crespo A, Verdu J, Ronda E. A reliable and valid questionnaire was developed to measure computer vision syndrome at the workplace. J Clin Epidemiol. 2015 Jun;68(6):662-73. doi: 10.1016/j.jclinepi.2015.01.015. Epub 2015 Jan 28. PMID 25744132